CLINICAL TRIAL: NCT01390207
Title: Does Earlier Administration Of Human Chorionic Gonadotropin (hCG) Improve The Probability Of Pregnancy In Cycles Stimulated With Rec-FSH AND GnRH Antagonists? A Prospective Randomized Trial
Brief Title: Earlier Triggering in Rec-FSH/GnRH Antagonist Cycles
Acronym: 16mm
Status: Completed | Phase: Phase 2 / Phase 3 | Type: Interventional
Sponsor: Universitair Ziekenhuis Brussel (Other)
Responsible Party: Kyrou Dimitra, Center of reproductive medicine-UZ
Allocation: Randomized | Model: Parallel | Masking: Double | Purpose: Treatment
Other Study IDs: 1971
Record Dates: First submitted 2011-05-19; First posted 2011-07-08 (Estimated); Last update posted 2011-08-04 (Estimated); Status verified 2011-07

CONDITIONS: hCG
Keywords: hCG triggering; pregnancy; GnRH antagonist

STUDY DESIGN:
Who Masked: Participant, Investigator
Oversight: Data Monitoring Committee: No

ARMS (1):
- 16mm follicles (Experimental)
  Interventions: Other: 16mm triggering

INTERVENTIONS:
Other: 16mm triggering — Final oocyte maturation will be achieved by administration of 10.000 IU of hCG (Pregnyl®). Randomization will be into 2 groups:
  • Group A (early hCG group): hCG will be administrated as soon as ≥ 3 follicles ≥ 16mm were present on ultrasound.

SUMMARY:
The effect of altering the timing of hCG administration on the ongoing pregnancy rate in patients stimulated with recombinant-FSH (rec-FSH)/gonadotrophin releasing hormone (GnRH) antagonists for in vitro fertilisation (IVF).

DETAILED DESCRIPTION:
Progesterone elevation has been associated with prolongation of the follicular phase in GnRH antagonists cycles by two days after the commonly used criterion of the presence of at least three follicles of >or= 17 mm has been met. Such an intervention is associated with significantly lower ongoing pregnancy rates in GnRH antagonist cycles, without an apparent deterioration of embryo quality.

The adverse effect of P elevation on the day of hCG administration might be explained by the induction of differences at the histological level as well as at the gene expression level between endometrial samples exposed to varying concentrations of progesterone (P). Prolongation of follicular phase by delaying hCG administration for two days is associated with a higher incidence of endometrial advancement on the day of oocyte retrieval in GnRH antagonist cycles (Kolibianakis et al., 2005). Moreover, Vaerenbergh et al., (2011) demonstrated a distinct difference in endometrial gene expression profile between patients with progesterone serum concentration above and below the threshold of 1.5 ng/ml on the day of HCG administration.

Due to the fact that earlier triggering of final oocyte maturation is expected to result in lower progesterone levels on the day of hCG administration it might be assumed that such an intervention might result in an improved probability of pregnancy by leading to a less deranged and more receptive endometrium.

The purpose of this randomized controlled trial is to evaluate whether triggering of final oocyte maturation as soon as ≥ 3 follicles ≥ 16mm are present on ultrasound or one day later affects the probability of pregnancy in patients stimulated with rec-FSH/GnRH- antagonists for IVF.

ELIGIBILITY:
Inclusion Criteria:- Age ≤ 39 years

* Body mass index between 18 and 29 kg/m²¬
* Presence of both ovaries
* Basal levels of estradiol (≤ 80 pg/ml) and progesterone (≤ 1.6ng/ml) on day one of the cycle
* Treatment with IVF/ICSI
* Embryo transfer on day 3 (1 or 2 embryos)
* Patients can enter in the study only once

Exclusion Criteria:

* Presence of endometriosis stage ≥3(AFS)
* Polycystic ovarian syndrome (Rotterdam criteria)
* Need for preimplantation genetic diagnosis (PGD)
* Azoospermia testicular sperm extraction (TESE)

Ages: 18 Years to 39 Years | Sex: Female | Healthy Volunteers: Yes
Age Groups: Adult
Enrollment: 100 (Actual)
Dates: Start 2010-01; Primary Completion 2011-04 (Actual); Study Completion 2011-05 (Actual)

PRIMARY OUTCOMES:
Ongoing pregnancy rate. | 1 year

SECONDARY OUTCOMES:
number of MII oocytes. | 1 year